CLINICAL TRIAL: NCT00709852
Title: A Multicenter, Randomized, Double-blind, Crossover, Phase 3 Study to Determine the Safety and Efficacy of Gadobutrol 1.0 Molar (Gadavist) in Patients Referred for Contrast-enhanced MRI of the Central Nervous System (CNS)
Brief Title: Safety and Efficacy of Gadobutrol 1.0 Molar (Gadavist) in Patients for Central Nervous System (CNS) Imaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 91681; 2007-004746-33 (EudraCT Number); 310123 (Other: Company Internal)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Diagnostic Imaging; Central Nervous System Diseases
Keywords: Patients referred for a contrast-enhanced MRI of the CNS; CNS Imaging
MeSH Terms: conditions — Central Nervous System Diseases | interventions — gadobutrol; gadoteridol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gadobutrol then Gadoteridol (Experimental): Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous) in Period 1 and a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. in Period 2.
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875); Drug: Gadoteridol (ProHance)
- Gadoteridol then Gadobutrol (Experimental): Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. in Period 1 and a single dose of gadobutrol 0.1 mmol/kg bw via i.v. in Period 2.
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875); Drug: Gadoteridol (ProHance)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous)
Drug: Gadoteridol (ProHance) — Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v.

SUMMARY:
This study involves the use of Magnetic Resonance Imaging (MRI) contrast agents called gadobutrol (Gadavist) Injection and ProHance Injection. The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of gadobutrol when used for taking MR images of the brain and spine. The results of the MRI with gadobutrol Injection will be compared to the results of MR images taken without contrast and with the results of the MR images taken with ProHance.

DETAILED DESCRIPTION:
Issues on safety will be addressed in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Is referred for a contrast-enhanced MRI of the CNS based on current clinical symptoms or results of a previous imaging procedure
* Has been fully informed about the study, including provisions of the Health Insurance Portability and Accountability Act (HIPAA) as applicable, and has consented to participate

Exclusion Criteria:

* Has any contraindication to the MRI examinations or the use of Gd-containing contrast agents
* Has a history of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents
* Has severe cardiovascular disease (eg, known long QT syndrome, acute myocardial infarction [< 14 days], unstable angina, congestive heart failure New York Heart Association class IV) or acute stroke (< 48 hours)- Patients with acute renal insufficiency of any severity due to hepato-renal syndrome or in the perioperative liver transplantation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (79):
- United States (24):
  - West Alabama Research, Inc., Birmingham, Alabama
  - Achieve Clinical Research, LLC, Tuscaloosa, Alabama
  - Los Gatos MRI, Los Gatos, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Redwood Regional Medical Group, Inc., Santa Rosa, California
  - University of Florida - Jacksonville, Jacksonville, Florida
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Atchison Hospital, Atchison, Kansas
  - University of Maryland Hospital System, Baltimore, Maryland
  - Johns Hopkins Hospital/Health System, Baltimore, Maryland
  - Shields MRI - Brockton, Brockton, Massachusetts
  - VA Boston Healthcare System-West Roxbury Division, West Roxbury, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Kingston Neurological Associates, PC, Kingston, New York
  - NYU Hospital for Joint Diseases, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- Austria (4):
  - Landeskrankenhaus Donauregion Tulln, Tulln, Lower Austria
  - Medizinische Universität Graz, Graz, Styria
  - LNK Wagner Jauregg, Linz, Upper Austria
  - Allgemeines Krankenhaus der Stadt Wien Universitätskliniken, Vienna, Vienna
- Colombia (4):
  - Fundación Instituto de Alta tecnología médica de Antioquia, Medellín, Antioquia
  - Fundación Santa Fe de Bogotá - Hospital Universitario, Bogotá, Cundinamarca
  - DIME Clinica Neurocardiovascular S.A., Cali, Valle del Cauca Department
  - Centro de Diagnostico Medico, Medellín
- Germany (20):
  - Deutsches Krebsforschungszentrum, Heidelberg, Baden-Wurttemberg
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe, Baden-Wurttemberg
  - Klinikum Mannheim gGmbH, Mannheim, Baden-Wurttemberg
  - Zentralklinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - LMU Klinikum der Universität München - Großhadern, München, Bavaria
  - Klinikum rechts der Isar, München, Bavaria
  - Klinikum Ernst von Bergmann, Potsdam, Brandenburg
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg, Hamburg
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Kliniken der Medizinischen Hochschule Hannover, Hanover, Lower Saxony
  - Medizinische Einrichtungen der Universität Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum Prof. Dr. D. Uhlenbrock, Dortmund, North Rhine-Westphalia
  - Universitätskliniken des Saarlandes, Homburg, Saarland
  - Medizinische Fakultät Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Klinikum der Christian-Albrechts-Universität, Kiel, Schleswig-Holstein
  - Universitätsklinikum Charite zu Berlin, Berlin, State of Berlin
  - HELIOS Klinikum Erfurt GmbH, Erfurt, Thuringia
- India (4):
  - CT /MRI centre, Indore, Madhya Pradesh
  - Piramal Diagnostic- Jankharia Imaging, Mumbai, Maharashtra
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Bombay Hospital, Institute of Medical sciences, Mumbai
- Japan (14):
  - Nagoya Kyoritsu Clinic, Nagoya, Aichi-ken
  - Nagoya Kyoritsu Hospital, Nagoya, Aichi-ken
  - Social Insurance Chukyo Hospital, Nagoya, Aichi-ken
  - Himeji Medical Center, Himeji, Hyōgo
  - Himeji Central Hospital, Himeji, Hyōgo
  - Institute of Biomedical Research and Innovation, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Shinsuma Hospital, Kobe, Hyōgo
  - Utano National Hospital, Kyoto, Kyoto
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka
  - Osaka National Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Shimonoseki Kosei Hospital, Shimonoseki, Yamaguchi
- Switzerland (5):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Hôpital Cantonal Universitaire de Genève, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of the first participant's first visit was 11 JUN 2008. The date of the last participant's last visit was 03 APR 2009.
Pre-assignment Details: A total of 419 participants (part.) were screened; 17 prematurely discontinued prior to receiving any study drug. A total of 402 part. received study drug; 228 in gadobutrol : gadoteridol treatment sequence, 174 in gadoteridol : gadobutrol treatment sequence. Safety analysis set=402; gadobutrol=399, gadoteridol=393. Full analysis set (FAS)=336.
Groups:
- Gadobutrol (Gadavist, BAY86-4875) : Gadoteridol (ProHance): Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous) in Period 1 and a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. in Period 2.
- Gadoteridol (ProHance) : Gadobutrol (Gadavist, BAY86-4875): Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. in Period 1 and a single dose of gadobutrol 0.1 mmol/kg bw via i.v. in Period 2.
Period: Period 1
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) : Gadoteridol (ProHance) | Gadoteridol (ProHance) : Gadobutrol (Gadavist, BAY86-4875)
Started | 228 | 174
Completed | 220 | 171
Not Completed | 8 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Defective scanner | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) : Gadoteridol (ProHance) | Gadoteridol (ProHance) : Gadobutrol (Gadavist, BAY86-4875)
Started | 220 | 171
Completed | 211 | 169
Not Completed | 9 | 2
Not completed — Protocol Violation | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — No 72-hour follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants who received either treatment
Arm/Group | Entire Study Population
Number analyzed (Participants) | 402
Age, Customized [Number; unit: participants]
  < 45 years | 144
  45-64 years | 164
  ≥ 65 years | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227
  Male | 175
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 235
  Black | 23
  Hispanic | 31
  Asian | 112
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: BR1 evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: The full analysis set (FAS); which used data from all participants for whom data and images were available for the unenhanced MRI, combined unenhanced and gadobutrol-enhanced MRI, and combined unenhanced and gadoteridol-enhanced MRI, excluding the sample participants (the first participant from each study site).
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Unenhanced: Participants had diagnostic imaging before receiving any contrast agent
- Combined Unenhanced/Gadobutrol-enhanced: Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous)
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 314 | 314
scores on a scale
  contrast enhancement | 0.94 (0.14) | 2.21 (0.57)
  border delineation | 2.03 (0.37) | 2.70 (0.53)
  internal morphology | 1.16 (0.26) | 1.78 (0.44)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.26, Standard Deviation 0.61
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t-test — for border delineation; Mean Difference (Final Values) = 0.67, Standard Deviation 0.66
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t-test — for internal morphology; Mean Difference (Final Values) = 0.62, Standard Deviation 0.47

2. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: BR2 evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 314 | 314
scores on a scale
  contrast enhancement | 1.01 (0.28) | 2.60 (0.70)
  border delineation | 2.19 (0.49) | 2.91 (0.60)
  internal morphology | 1.46 (0.37) | 2.28 (0.47)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.59, Standard Deviation 0.77
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Median Difference (Final Values) = 0.72, Standard Deviation 0.78
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.82, Standard Deviation 0.61

3. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: BR3 evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 312 | 312
scores on a scale
  contrast enhancement | 0.96 (0.16) | 2.02 (0.46)
  border delineation | 1.73 (0.32) | 2.16 (0.35)
  internal morphology | 1.34 (0.32) | 1.76 (0.39)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.06, Standard Deviation 0.51
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.43, Standard Deviation 0.50
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.41, Standard Deviation 0.52

4. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Average Reader (AR)
Description: The AR analysis used the mean of the values for the 3 blinded readers. The 3 BRs evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 316 | 316
scores on a scale
  contrast enhancement | 0.97 (0.15) | 2.26 (0.52)
  border delineation | 1.98 (0.30) | 2.58 (0.43)
  internal morphology | 1.32 (0.24) | 1.93 (0.36)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.29, Standard Deviation 0.56
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.60, Standard Deviation 0.53
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.61, Standard Deviation 0.42

5. Primary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Readers
Description: The blinded readers evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 336 | 336
lesions
  BR1 | 7.41 (13.05) | 7.80 (12.92)
  BR2 | 10.07 (16.60) | 9.63 (15.04)
  BR3 | 6.75 (8.97) | 7.31 (9.13)
  AR | 8.08 (12.39) | 8.25 (11.40)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; BR 1; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.199 to 0.984], Standard Deviation 5.51
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; BR 2; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval (CI) is compared to noninferiority margin; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.772 to 0.885], Standard Deviation 12.38
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; BR 3; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.125 to 1.000], Standard Deviation 4.07
Statistical Analysis 4: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; AR; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.439 to 0.780], Standard Deviation 5.68

6. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: as for outcome 1
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  contrast enhancement | 1.00 (0.04) | 2.62 (0.30)
  border delineation | 2.14 (0.21) | 2.95 (0.31)
  internal morphology | 1.26 (0.22) | 2.03 (0.33)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.62, Standard Deviation 0.30
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.81, Standard Deviation 0.37
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.77, Standard Deviation 0.38

7. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: as for outcome 2
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  contrast enhancement | 1.15 (0.45) | 3.28 (0.40)
  border delineation | 2.36 (0.33) | 3.22 (0.37)
  internal morphology | 1.44 (0.31) | 2.54 (0.27)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 2.13, Standard Deviation 0.62
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.86, Standard Deviation 0.46
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 1.10, Standard Deviation 0.39

8. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: as for outcome 3
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  contrast enhancement | 1.04 (0.14) | 2.39 (0.29)
  border delineation | 1.75 (0.20) | 2.25 (0.28)
  internal morphology | 1.42 (0.21) | 1.85 (0.26)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.36, Standard Deviation 0.33
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.50, Standard Deviation 0.33
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.43, Standard Deviation 0.32

9. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader (AR)
Description: as for outcome 4
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  contrast enhancement | 1.06 (0.16) | 2.76 (0.23)
  border delineation | 2.09 (0.17) | 2.81 (0.21)
  internal morphology | 1.38 (0.16) | 2.14 (0.18)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.70, Standard Deviation 0.30
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.72, Standard Deviation 0.23
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.76, Standard Deviation 0.22

10. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: as for outcome 1
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 267 | 267
scores on a scale
  contrast enhancement | 0.86 (0.30) | 1.69 (1.04)
  border delineation | 1.89 (0.74) | 2.40 (0.94)
  internal morphology | 1.04 (0.47) | 1.48 (0.74)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 0.83, Standard Deviation 1.16
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.52, Standard Deviation 1.26
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.44, Standard Deviation 0.82

11. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: as for outcome 2
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 274 | 274
scores on a scale
  contrast enhancement | 0.87 (0.31) | 1.75 (1.17)
  border delineation | 1.97 (0.83) | 2.51 (1.06)
  internal morphology | 1.47 (0.67) | 1.95 (0.83)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 0.89, Standard Deviation 1.29
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.54, Standard Deviation 1.44
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.48, Standard Deviation 1.11

12. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: as for outcome 3
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 277 | 277
scores on a scale
  contrast enhancement | 0.86 (0.30) | 1.55 (0.83)
  border delineation | 1.72 (0.63) | 2.05 (0.63)
  internal morphology | 1.26 (0.60) | 1.64 (0.70)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 0.69, Standard Deviation 0.95
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.33, Standard Deviation 0.97
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.39, Standard Deviation 0.96

13. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader (AR)
Description: as for outcome 4
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 293 | 293
scores on a scale
  contrast enhancement | 0.85 (0.26) | 1.62 (0.95)
  border delineation | 1.82 (0.62) | 2.26 (0.81)
  internal morphology | 1.23 (0.47) | 1.65 (0.66)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 0.78, Standard Deviation 1.06
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.44, Standard Deviation 1.07
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.42, Standard Deviation 0.83

14. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Average Reader
Description: as for outcome 4
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Combined Unenhanced/Gadoteridol-enhanced: Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v.
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 315 | 315
scores on a scale
  contrast enhancement | 0.98 (0.14) | 2.22 (0.50)
  border delineation | 1.99 (0.28) | 2.55 (0.41)
  internal morphology | 1.32 (0.22) | 1.90 (0.35)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for contrast enhancement; Mean Difference (Final Values) = 1.24, Standard Deviation 0.53
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.56, Standard Deviation 0.48
Statistical Analysis 3: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.58, Standard Deviation 0.41

15. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Average Reader
Description: The AR analysis used the mean of the values for the 3 blinded readers
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 8.08 (12.39) | 8.24 (11.79)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.532 to 0.851], Standard Deviation 6.44

16. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Average Reader
Description: The AR analysis used the mean of the values for the 3 blinded readers.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Combined Unenhanced/Gadobutrol-enhanced: Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v.
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 315 | 315
scores on a scale
  contrast enhancement | 2.28 (0.51) | 2.24 (0.49)
  border delineation | 2.60 (0.39) | 2.56 (0.39)
  internal morphology | 1.94 (0.34) | 1.91 (0.34)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for contrast enhancement; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.04, 95% CI [0.0004 to 0.078], Standard Deviation 0.33
Statistical Analysis 2: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for border delineation; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.04, 95% CI [-0.009 to 0.082], Standard Deviation 0.41
Statistical Analysis 3: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for internal morphology; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.03, 95% CI [-0.006 to 0.059], Standard Deviation 0.29

17. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Average Reader
Description: The AR analysis used the mean of the values for the 3 blinded readers
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 8.25 (11.40) | 8.24 (11.79)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.01, 95% CI [-0.601 to 0.622], Standard Deviation 5.70

18. Secondary Outcome: Percentage of Participants With More Lesions Detected for Combined Unenhanced/Gadobutrol-enhanced MRI or for Unenhanced MRI by Blinded Readers
Description: The AR analysis used the mean of the values for the 3 blinded readers. The 3 BRs evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another and determined the number of lesion from each.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced: Participants had diagnostic imaging before receiving any contrast agent. Lesions detected by Unenhanced MRI were compared to Combined Unenhanced/Gadobutrol-enhanced MRI.
- Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced: Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous). Lesions detected by Combined Unenhanced/Gadobutrol-enhanced MRI were compared to Unenhanced MRI.
Arm/Group | Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced
Number analyzed (Participants) | 336 | 336
percentage of participants
  BR1 | 26.5 | 34.8
  BR2 | 35.4 | 34.5
  BR3 | 24.4 | 40.2
  AR | 35.1 | 44.0
Statistical Analysis 1: Comparison: Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced; Test type: Superiority or Other; Difference in percentages = 8.3 — for BR1
Statistical Analysis 2: Comparison: Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced; Test type: Superiority or Other; Difference in percentages = -0.9 — for BR2
Statistical Analysis 3: Comparison: Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced; Test type: Superiority or Other; Difference in percentages = 15.8 — for BR3
Statistical Analysis 4: Comparison: Unenhanced Compared to Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadobutrol-enhanced Compared to Unenhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; confidence interval is given for AR; lower limit is compared to the noninferiority margin; Difference in percentages = 8.9, 95% CI 2-sided [-0.5 to 18.4]

19. Secondary Outcome: Percentage of Participants With More Lesions Detected for Combined Unenhanced/Gadoteridol-enhanced MRI or for Unenhanced MRI by Average Reader
Description: The AR analysis used the mean of the values for the 3 blinded readers. The 3 BRs evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadoteridol-enhanced MRIs in another and determined the number of lesion from each.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Unenhanced Compared to Gadoteridol-enhanced: Participants had diagnostic imaging before receiving any contrast agent. Lesions detected by Unenhanced MRI were compared to Combined Unenhanced/Gadoteridol-enhanced MRI.
- Gadoteridol-enhanced Compared to Unenhanced: Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. Lesions detected by Combined Unenhanced/Gadoteridol-enhanced MRI were compared to Unenhanced MRI.
Arm/Group | Unenhanced Compared to Gadoteridol-enhanced | Gadoteridol-enhanced Compared to Unenhanced
Number analyzed (Participants) | 336 | 336
percentage of participants | 37.8 | 41.4
Statistical Analysis 1: Comparison: Unenhanced Compared to Gadoteridol-enhanced vs Gadoteridol-enhanced Compared to Unenhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 3.6, 95% CI [-5.9 to 13.1]

20. Secondary Outcome: Percentage of Participants With More Lesions Detected for Combined Unenhanced/Gadobutrol-enhanced MRI or for Combined Unenhanced/Gadoteridol-enhanced MRI by Average Reader
Description: The AR analysis used the mean of the values for the 3 blinded readers. The 3 BRs evaluated the images from the combined unenhanced and gadobutrol-enhanced MRIs in one session and the images from the combined unenhanced and gadoteridol-enhanced MRIs in another and determined the number of lesion from each.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Gadobutrol-enhanced Compared to Gadoteridol-enhanced: Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. Lesions detected by Combined Unenhanced/Gadobutrol-enhanced MRI were compared to Combined Unenhanced/Gadoteridol-enhanced MRI.
- Gadoteridol-enhanced Compared to Gadobutrol-enhanced: Participants received a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v. Lesions detected by Combined Unenhanced/Gadoteridol-enhanced MRI were compared to Combined Unenhanced/Gadobutrol-enhanced MRI.
Arm/Group | Gadobutrol-enhanced Compared to Gadoteridol-enhanced | Gadoteridol-enhanced Compared to Gadobutrol-enhanced
Number analyzed (Participants) | 336 | 336
percentage of participants | 41.7 | 33.3
Statistical Analysis 1: Comparison: Gadobutrol-enhanced Compared to Gadoteridol-enhanced vs Gadoteridol-enhanced Compared to Gadobutrol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 8.3, 95% CI [-0.9 to 17.6]

21. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI and the images from the combined unenhanced and gadobutrol-enhanced MRIs. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 329 | 329
scores on a scale
  border delineation | 2.16 (0.62) | 2.90 (0.62)
  internal morphology | 1.77 (0.55) | 2.38 (0.50)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.74, Standard Deviation 0.78
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.61, Standard Deviation 0.61

22. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 3.46 (7.99) | 3.75 (8.09)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.29, 95% CI [-0.053 to 0.636], Standard Deviation 3.21

23. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: as for outcome 21
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  border delineation | 2.13 (0.55) | 2.90 (0.54)
  internal morphology | 1.76 (0.48) | 2.40 (0.44)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.77, Standard Deviation 0.64
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.64, Standard Deviation 0.50

24. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: as for outcome 21
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 272 | 272
scores on a scale
  border delineation | 2.20 (0.95) | 2.94 (0.99)
  internal morphology | 1.80 (0.80) | 2.36 (0.76)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.74, Standard Deviation 1.26
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.56, Standard Deviation 0.97

25. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI and the images from the combined unenhanced and gadoteridol-enhanced MRIs. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 329 | 329
scores on a scale
  border delineation | 2.17 (0.61) | 2.88 (0.60)
  internal morphology | 1.78 (0.55) | 2.36 (0.49)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.71, Standard Deviation 0.76
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.58, Standard Deviation 0.63

26. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI and the images from the combined unenhanced and gadoteridol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 3.46 (7.99) | 3.74 (8.15)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.28, 95% CI [-0.087 to 0.641], Standard Deviation 3.39

27. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: as for outcome 25
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  border delineation | 2.13 (0.55) | 2.91 (0.52)
  internal morphology | 1.76 (0.48) | 2.39 (0.43)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.78, Standard Deviation 0.61
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.63, Standard Deviation 0.49

28. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: as for outcome 25
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 270 | 270
scores on a scale
  border delineation | 2.23 (0.94) | 2.88 (0.97)
  internal morphology | 1.83 (0.79) | 2.34 (0.77)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.65, Standard Deviation 1.27
Statistical Analysis 2: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.51, Standard Deviation 1.01

29. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the combined unenhanced and gadobutrol-enhanced MRIs and the images from the combined unenhanced and gadoteridol-enhanced MRIs. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 328 | 328
scores on a scale
  contrast enhancement | 2.67 (0.70) | 2.60 (0.72)
  border delineation | 2.95 (0.55) | 2.91 (0.56)
  internal morphology | 2.42 (0.45) | 2.39 (0.46)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for contrast enhancement; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.06, 95% CI [0.030 to 0.096]
Statistical Analysis 2: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for border delineation; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.04, 95% CI [0.003 to 0.071]
Statistical Analysis 3: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for internal morphology; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.03, 95% CI [0.003 to 0.055]

30. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the combined unenhanced and gadobutrol-enhanced MRIs and the combined unenhanced and gadoteridol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 3.75 (8.09) | 3.74 (8.15)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; confidence interval for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.01, 95% CI [-0.049 to 0.078], Standard Deviation 0.59

31. Secondary Outcome: Scores for Contrast Enhancement, Border Delineation and Internal Morphology for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: as for outcome 29
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 310 | 310
scores on a scale
  contrast enhancement - gadobutrol combined | 2.88 (0.52) | 2.85 (0.54)
  border delineation - gadobutrol combined | 2.90 (0.54) | 2.91 (0.52)
  internal morphology - gadobutrol combined | 2.40 (0.44) | 2.39 (0.43)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for contrast enhancement; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.03, 95% CI [-0.009 to 0.065]
Statistical Analysis 2: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for border delineation; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = -0.01, 95% CI [-0.040 to 0.020]
Statistical Analysis 3: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for internal morphology; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.01, 95% CI [-0.015 to 0.035]

32. Secondary Outcome: Scores for Contrast Enhancement, Border Delineation and Internal Morphology for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: as for outcome 29
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 263 | 263
scores on a scale
  contrast enhancement | 2.44 (1.21) | 2.34 (1.22)
  border delineation | 3.04 (0.88) | 2.94 (0.84)
  internal morphology | 2.44 (0.63) | 2.39 (0.69)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for contrast enhancement; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.10, 95% CI [0.042 to 0.153]
Statistical Analysis 2: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for border delineation; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.10, 95% CI [0.030 to 0.161]
Statistical Analysis 3: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; analysis for internal morphology; Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; CI for paired means; lower limit of confidence interval is compared to noninferiority margin; Mean Difference (Final Values) = 0.05, 95% CI [0.006 to 0.098]

33. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the BRs. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the majority reader diagnoses for the combined unenhanced/gadobutrol-enhanced and the unenhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 225 | 225
per. of the exact diagnostic matches | 58.2 | 64.4
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.0082, McNemar; Difference = 6.2

34. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the investigator diagnoses for the combined unenhanced/gadobutrol-enhanced and the unenhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 292 | 292
per. of the exact diagnostic matches | 69.2 | 79.1
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 9.9

35. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the BRs. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the majority reader diagnoses for the combined unenhanced/gadoteridol-enhanced and the unenhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 219 | 219
per. of the exact diagnostic matches | 58.9 | 65.8
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.0039, McNemar; Difference = 6.8

36. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the investigator diagnoses for the combined unenhanced/gadoteridol-enhanced and the unenhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
per. of the exact diagnostic matches | 69.2 | 78.4
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 9.2

37. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the BRs. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the majority reader diagnoses for the combined unenhanced/gadobutrol-enhanced and the combined unenhanced/gadoteridol-enhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 229 | 229
per. of the exact diagnostic matches | 65.1 | 65.5
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = -0.4, 95% CI [-3.8 to 2.9]

38. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the clinical investigator diagnoses for the combined unenhanced/gadobutrol-enhanced and the combined unenhanced/gadoteridol-enhanced MR images were evaluated for consistency with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
per. of the exact diagnostic matches | 79.1 | 78.4
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of interval is compared to noninferiority margin; Difference in percentages = 0.7, 95% CI [-0.3 to 1.6]

39. Secondary Outcome: Accuracy of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of abnormal brain tissue.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 267 | 267
percentage of participants | 66.7 | 77.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.0002, McNemar; Difference = 10.5

40. Secondary Outcome: Sensitivity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 206 | 206
percentage of participants | 62.6 | 76.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 13.6

41. Secondary Outcome: Specificity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 61 | 61
percentage of participants | 80.3 | 80.3
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 1.0000, McNemar; Difference = 0.0

42. Secondary Outcome: Accuracy of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of abnormal brain tissue.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 267 | 267
percentage of participants | 66.7 | 77.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.0002, McNemar; Difference = 10.5

43. Secondary Outcome: Sensitivity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly detects abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 206 | 206
percentage of participants | 62.6 | 75.7
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.0001, McNemar; Difference = 13.1

44. Secondary Outcome: Specificity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly excludes abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 61 | 61
percentage of participants | 80.3 | 82.0
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.7630, McNemar; Difference = 1.6

45. Secondary Outcome: Accuracy of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of abnormal brain tissue.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 267 | 267
percentage of participants | 77.2 | 77.2
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 0.0, 95% CI [-3.1 to 3.1]

46. Secondary Outcome: Sensitivity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly detects abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 206 | 206
percentage of participants | 76.2 | 75.7
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 0.5, 95% CI [-2.7 to 3.6]

47. Secondary Outcome: Specificity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly excludes abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 61 | 61
percentage of participants | 80.3 | 82.0
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = -1.6, 95% CI [-10.1 to 6.9]

48. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 81.2 | 87.7
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.0006, McNemar; Difference = 6.5

49. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 47.3 | 66.7
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.0004, McNemar; Difference = 19.4

50. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 97.0 | 97.5
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.6547, McNemar; Difference = 0.5

51. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 87.3 | 95.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 7.9

52. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 66.7 | 88.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 21.5

53. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 97.0 | 98.5
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p = 0.0833, McNemar; Difference = 1.5

54. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 81.2 | 85.6
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.0236, McNemar; Difference = 4.5

55. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly detects malignant lesions as defined by the independent truth committee
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 47.3 | 60.2
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.0186, McNemar; Difference = 12.9

56. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 97.0 | 97.5
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.7055, McNemar; Difference = 0.5

57. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 87.3 | 94.5
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 7.2

58. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 66.7 | 87.1
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, McNemar; Difference = 20.4

59. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadoteridol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 97.0 | 98.0
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p = 0.1573, McNemar; Difference = 1.0

60. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 87.7 | 85.6
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 2.1, 95% CI [0.2 to 3.9]

61. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 66.7 | 60.2
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 6.5, 95% CI [1.5 to 11.4]

62. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 97.5 | 97.5
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 0.0, 95% CI [-1.4 to 1.4]

63. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 292 | 292
percentage of participants | 95.2 | 94.5
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 0.7, 95% CI [-0.3 to 1.6]

64. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 93 | 93
percentage of participants | 88.2 | 87.1
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 1.1, 95% CI [-1.0 to 3.2]

65. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (Gadobutrol-enhanced or Gadoteridol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 199 | 199
percentage of participants | 98.5 | 98.0
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Non-Inferiority or Equivalence — noninferiority margin = -10%; CI for paired percentages; lower limit of confidence interval is compared to noninferiority margin; Difference in percentages = 0.5, 95% CI [-0.5 to 1.5]

66. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader
Description: The BRs recorded his/her confidence in diagnosis for the unenhanced MR image set and the combined unenhanced/enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident. The AR score was the mean of the means of the 3 BRs.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 2.23 (0.48) | 2.80 (0.54)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test; Mean Difference (Final Values) = 0.57, Standard Deviation 0.56

67. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Average Reader
Description: as for outcome 66
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 2.23 (0.48) | 2.80 (0.54)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test; Mean Difference (Final Values) = 0.57, Standard Deviation 0.58

68. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Average Reader
Description: The BRs recorded his/her confidence in diagnosis for the combined unenhanced/enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident. The AR score was the mean of the means of the 3 BRs.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 2.80 (0.54) | 2.80 (0.54)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, Standard Deviation 0.48

69. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The investigator recorded his/her confidence in diagnosis for the unenhanced MR image set and the combined unenhanced/gadobutrol-enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadobutrol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 2.59 (1.02) | 3.35 (0.76)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadobutrol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test; Mean Difference (Final Values) = 0.76, Standard Deviation 0.93

70. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadoteridol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The investigator recorded his/her confidence in diagnosis for the unenhanced MR image set and the combined unenhanced/gadoteridol-enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident.
Time Frame: Up to 2 hours after injection of gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 2.59 (1.02) | 3.31 (0.79)
Statistical Analysis 1: Comparison: Unenhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; p < 0.0001, paired t test; Mean Difference (Final Values) = 0.73, Standard Deviation 0.89

71. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Combined Unenhanced/Gadoteridol-enhanced MRI by Clinical Investigator
Description: The investigator recorded his/her confidence in diagnosis for the combined unenhanced/gadobutrol-enhanced MR image sets and the combined unenhanced/gadoteridol MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
scores on a scale | 3.35 (0.76) | 3.31 (0.79)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; Mean Difference (Final Values) = 0.04, Standard Deviation 0.39

72. Secondary Outcome: Comparison of Image Quality Between Gadobutrol and Gadoteridol by Blinded Readers
Description: The BRs evaluated the relative image quality of the gadobutrol-enhanced T1w MR images and the gadoteridol-enhanced T1w MR images in a paired fashion on a 5-point scale where 1 = image on right was worse, 2 = image on right was slightly worse, 3 = both images were the same, 4 = image on right was slightly better, and 5 = image on right was better.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Combined Gadobutrol vs. Combined Gadoteridol: Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous) and a single dose of gadoteridol at the approved dose, 0.1 mmol/kg bw, via i.v.
Arm/Group | Combined Gadobutrol vs. Combined Gadoteridol
Number analyzed (Participants) | 336
scores on a scale
  blinded reader 4 | 0.33 (0.78)
  blinded reader 5 | 0.38 (0.83)
  blinded reader 6 | 0.53 (1.24)
Statistical Analysis 1: Comparison: Combined Gadobutrol vs. Combined Gadoteridol; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — for all three readers

73. Secondary Outcome: Percentage of Participants for Which Blinded Readers Said Image Quality Was Higher
Description: Percentage of participants for which blinded readers said image quality was higher
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
percentage of participants
  BR 4 | 36.0 | 7.5
  BR 5 | 35.1 | 7.5
  BR 6 | 62.2 | 24.4

74. Secondary Outcome: Assessment of the Number of Contrast-enhanced Lesions for Gadobutrol and Gadoteridol by Blinded Readers
Description: Two BRs independently provided the number of contrast-enhanced lesions for gadobutrol and gadoteridol. In cases of disagreement between the readers, an independent adjudicator provided the number of contrast-enhanced lesions. The adjudicator results were used in the analysis in the cases of disagreement between the original readers
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 336 | 336
lesions | 1.73 (4.74) | 1.73 (4.89)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, Standard Deviation 1.06

75. Secondary Outcome: Percentage of Lesion Enhancement From Unenhanced to Combined Unenhanced/Enhanced for Gadobutrol and Gadoteridol by Blinded Readers
Description: From the quantitative signal intensity values assessed by the BR, the percentage of lesion enhancement from unenhanced to combined unenhanced/enhanced was calculated.
Time Frame: Up to 2 hours after injection of gadobutrol or gadoteridol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of lesion enhancement
Arm/Group | Combined Unenhanced/Gadobutrol-enhanced | Combined Unenhanced/Gadoteridol-enhanced
Number analyzed (Participants) | 185 | 185
percentage of lesion enhancement | 80.1 (58.4) | 77.7 (52.3)
Statistical Analysis 1: Comparison: Combined Unenhanced/Gadobutrol-enhanced vs Combined Unenhanced/Gadoteridol-enhanced; Test type: Superiority or Other; Mean Difference (Final Values) = 2.4, Standard Deviation 26.6

ADVERSE EVENTS:
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Participants received a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous)
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadoteridol (ProHance)
Serious Adverse Events (participants affected / at risk) | 2/399 | 1/393
Other Adverse Events (participants affected / at risk) | 46/399 | 45/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=399) | Gadoteridol (ProHance) (N=393)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=399) | Gadoteridol (ProHance) (N=393)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Nausea (Gastrointestinal disorders) | 11 (11) | 17 (18)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 4 (4) | 1 (1)
Blood glucose increased (Investigations) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 5 (5)
Dysgeusia (Nervous system disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 13 (13) | 10 (12)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study it performs. All relevant aspects regarding publication will be part of the contract between the sponsor and the investigator/institution. The sponsor has committed to the global industry position on disclosure of information about clinical trials. The information regarding the study protocol is made publicly available on the internet at www.clinicaltrials.gov.